CLINICAL TRIAL: NCT06186505
Title: Heat Therapy for Peripheral Arterial Disease (HEATPAD)
Acronym: HEATPAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: GreenCross Medico Limited (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 304872 (42-03-21)
Record Dates: First submitted 2021-11-05; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication; Critical Limb Ischemia
Keywords: Healthy volunteers; AirGlove; Heat therapy; Walking distance
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Chronic Limb-Threatening Ischemia; Hyperthermia

STUDY DESIGN:
Intervention Model Description: All cohorts of study will receive heat therapy from AirGlove device. Patient cohorts will undergo 12 weeks of heat therapy. Healthy control cohort will only receive a single session of heat therapy.
Masking Description: By the nature of the study treatments used within this study, blinding of the participants and clinicians is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1a (Experimental): Phase 1a will be undertaken in 10 healthy volunteers to assess the effects of the AirGlove device on lower limb arterial flow, tissue perfusion, and product usability following a single session. Measurements will be taken just prior to device application, and then again at the time of device removal.
  Interventions: Device: AirGlove
- Phase 1b (Experimental): Phase 1b will be undertaken in 20 PAD patients with intermittent claudication to assess the effects of the AirGlove device on lower limb arterial flow, tissue perfusion, quality of life and product usability both in a single session, and following a 12-week trial of heat therapy. Measurements will be taken just prior to device application, and then again at the time of device removal at the start of the trial, and again at week 12 (in line with the recommended duration of SET).
  Interventions: Device: AirGlove
- Phase 1c (Experimental): Phase 1c will be undertaken in 10 PAD patients with critical limb ischaemia Rutherford stage 4 (rest pain). Lower limb arterial flow, tissue perfusion, pain scores, quality of life, and product usability will be assessed both in a single session and following a 2-12 week trial of heat therapy.
  Interventions: Device: AirGlove

INTERVENTIONS:
Device: AirGlove — AirGlove is a unique warming system developed to enable access to the veins in a patients arm for the delivery of intraveneous drugs by gently heating the patients arm up as it forces warm air through a double walled polythene glove. In this study, the device will be used on the leg of the participants as means of encouraging circulation to the area.
  Other Names: GB001

SUMMARY:
Peripheral arterial disease (PAD) is a disabling condition, with symptoms of muscle cramping or pain on exertion, which can substantially reduce quality of life. This study aims to see if AirGlove device improves participants circulation. This is phase 1 study and will be taken in 3 parts: Phase 1a will be undertaken in 10 healthy volunteers to assess the effects of the AirGlove device on lower limb arterial flow, tissue perfusion, quality of life and product usability following a single session. Phase 1b will be undertaken in 20 participants with intermittent claudication to assess the effects of the AirGlove device on lower limb arterial flow, tissue perfusion, quality of life and product usability both in a single session and following a 12-week trial of heat therapy. Phase 1c will be undertaken in 10 participants with critical limb ischaemia Rutherford stage 4 (rest pain). Lower limb arterial flow, tissue perfusion, pain scores, quality of life, and product usability will be assessed both in a single session and following a 2-12 week trial of heat therapy.

DETAILED DESCRIPTION:
As people get older, the blood supply to the legs can get worse. This is caused by blockages in the main blood vessels in the leg. If left to get worse this can progress to ulcers and amputation. If treated early the blood supply can be improved. Currently patients are advised to exercise to improve their blood supply, however not all patients can do this. Recent work has shown that heat treatment could have a benefit in these patients to help improve walking distance and lower the risk of amputation. The studies so far have been limited to a one-off treatment, typically to the whole body rather than the affected leg. This study aims to use a device to warm the lower leg for a set amount of timeper day. The research team will look at the improvement in their walking distance and blood supply to the leg over a 12 week period.

The first phase of this study will be in healthy volunteers. They will undergo the trial protocol in a single session to assess acceptability of the trial protocol and identify potential barriers.

All patients invited into this study will be given the heat therapy device called AirGlove. This slides over the lower leg like a large sock, and hot air circulates within the sock itself. The research team will teach the patient how to use the device and they will then take it home for 12 weeks. At the start and end of the study patients will undergo tests to assess their walking distance, quality of life, pain, and to assess how much blood is getting down their leg.

This study will look at the role of heat therapy as an alternative to help improve their walking, potentially reducing the need for surgery, and saving legs.

ELIGIBILITY:
Participants in Phase 1a will be healthy volunteers. The inclusion criteria for this cohort are:

* Aged 18 or over
* ABPI within normal range (0.9 - 1.2)
* Negative Edinburgh Claudication Questionnaire

For Phase 1b and 1c inclusion criteria are:

* Capacity to provide informed consent
* Aged 60 or over
* ABPI <0.9
* Positive Edinburgh Claudication Questionnaire

Exclusion Criteria:

* Aged under 60 years (for Phase 1b and 1c only)
* Has known allergy to any trial product
* undergone previous surgical or endovascular intervention for peripheral arterial or endovascular intervention for peripheral arterial disease
* Alternative cause of leg pain
* Requires urgent revascularisation (<2 weeks)
* Significant leg ulceration/necrosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in walking distance. | Participants in phases 1b and 1c will be measured at baseline and at a 12-week follow up visit. Participants in phase 1c will additionally have their walking distance measured at visits at 3 and 6 weeks.
  Participants in phase 1b and 1c will undergo a 6-minute walk test to measure the initial claudication distance and maximum claudication distance.

SECONDARY OUTCOMES:
Change in tissue perfusion. | Participants in phases 1b and 1c will be measured at baseline and at a 12-week follow up visit. Participants in phase 1c will additionally be measured at visits at 3 and 6 weeks.
  A laser doppler flowmeter will be used to measure change in tissue perfusion.
Change in arterial blood flow. | Participants in phases 1b and 1c will be measured at baseline and at a 12-week follow up visit. Participants in phase 1c will additionally be measured at visits at 3 and 6 weeks.
  A doppler ultrasound will be used to measure blood volume flow and time adjusted mean velocity in the common femoral artery. Blood volume flow compromises the volume of blood crossing a single point in the common femoral artery, whereas time adjusted mean velocity is the rate of change of blood flow at this point. These assessments will be undertaken prior to application of the AirGlove device, and just prior to device removal at 30 minutes. Further haemodynamic assessments will be undertaken 10 minutes, 20 minutes, and 30 minutes post device removal. This will be assessed in this manner during each participant visit.
Change in ankle brachial pressure index and toe pressure index. | Participants in phases 1b and 1c will be measured at baseline and at a 12-week follow up visit. Participants in phase 1c will additionally be measured at visits at 3 and 6 weeks.
  ABPI measurements will also be undertaken at the same timepoints both pre and post device removal. These assessments will be undertaken prior to application of the AirGlove device, and just prior to device removal at 30 minutes. Further haemodynamic assessments will be undertaken 10 minutes, 20 minutes, and 30 minutes post device removal.
EQ-5D-5L Questionnaire score | Participants in phases 1b and 1c will be measured at baseline and at a 12-week follow up visit. Participants in phase 1c will additionally be measured at visits at 3 and 6 weeks.
  Participants in phases 1b and 1c will complete the EQ-5D-5L questionnaire to assess quality of life.
Intermittent Claudication Questionnaire score | Participants in phases 1b and 1c will be measured at baseline and at a 12-week follow up visit. Participants in phase 1c will additionally be measured at visits at 3 and 6 weeks.
  Participants in phases 1b and 1c will complete the Intermittent Claudication Questionnaire to assess quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Stather, Mr, Principal Investigator — Norfolk and Norwich University Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No